CLINICAL TRIAL: NCT05448417
Title: Exploration of Non-invasive High-frequency Oscillations in Human-machine Asynchrony in Healthy Subjects : a Clinical Crossover Trial
Brief Title: Exploration of Non-invasive High-frequency Oscillations in Human-machine Asynchrony in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jianyi Niu, Principle investigator, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GZ-202203
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Non-invasive Ventilation; Healthy Subjects
Keywords: Noninvasive high frequency oscillatory ventilation

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive one hour each of the two non-invasive ventilation modes before and after, and one hour of washout after receiving the first mode of ventilation before receiving the second intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-invasive high-frequency oscillatory ventilation (Experimental): Patients were titrated for relevant parameters of noninvasive ventilation the day before the trial. In the non-invasive high-frequency oscillation ventilation mode, the support pressure is consistent with the noninvasive bi-level positive pressure mode, and the highfrequency airway pressure oscillation driven by the solenoid valve is added during the expiratory phase. The amplitude is about 4cmH2O, and the oscillation frequency is about 8HZ.
  Interventions: Device: Non-invasive high-frequency oscillatory ventilation
- Bilevel positive pressure ventilation (Active Comparator): Bilevel positive pressure ventilation Patients were titrated for relevant parameters of non-invasive ventilation the day before the trial. Noninvasive bilevel positive pressure ventilation mode pressure titration follows previous studies.
  Interventions: Device: Noninvasive Bilevel Positive Pressure Ventilation

INTERVENTIONS:
Device: Non-invasive high-frequency oscillatory ventilation — Non-invasive high-frequency oscillatory ventilation generates high-frequency pressure fluctuations in the airway caused by the opening and closing of a solenoid valve.
  Arms: non-invasive high-frequency oscillatory ventilation
Device: Noninvasive Bilevel Positive Pressure Ventilation — Noninvasive Bilevel Positive Pressure Ventilation
  Arms: Bilevel positive pressure ventilation

SUMMARY:
High-frequency oscillatory ventilation (HFOV), as an ideal lung-protecting ventilation method, has been gradually applied to neonatal intensive care treatment, and is currently recommended as a rescue method for neonatal acute respiratory distress syndrome (ARDS) after conventional mechanical treatment fails. ventilation. Non-invasive high-frequency oscillatory ventilation (nHFOV) combines the advantages of HFOV and non-invasive ventilation methods, and has become a research hotspot in this field. Recommended to avoid intubation after failure of conventional non-invasive ventilation therapy. There is a lack of large-scale clinical trials systematically exploring its efficacy for intubation therapy. The increasing clinical application of nHFOV has also enriched its application in the treatment of other diseases. Human-machine asynchrony during non-invasive ventilation will seriously affect its efficacy, but no one has reported on the research related to nHFOV human-machine asynchrony.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-40, males and females;
2. Pulmonary function test found that the subject's lung function was normal;
3. Pulmonary disease not related to the results of the experiment;
4. Willing to participate in the study;
5. Able to provide informed consent.

Exclusion Criteria:

1. Bronchiectasis; post-tuberculosis sequelae; rib cage deformities; neuromuscular disorders; and bronchial carcinoma.
2. Intolerant with NIV

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Asynchrony index | 1 hour
  Asynchrony index is defined as the number of asynchrony events divided by the total espiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts: asynchrony Index (expressed in percentage) = number of asynchrony events/total respiratory rate (ventilator cycles +wasted efforts) × 100

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangdong, China